CLINICAL TRIAL: NCT02434536
Title: Assessment of the Appropriateness Admission From Emergency Departments in the Exacerbation of COPD. Validity of Explicit Criteria and Study of the Variability Between Different Centers of NHS. Multicenter Study IRYSS-Appropriateness-COPD.
Brief Title: Appropriate Admission in COPD Exacerbation From Emergency Department. Multicenter Study
Acronym: IRYSS-COPD
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, JOSE M QUINTANA-LOPEZ, MD PhD, PhD, MD, Hospital Galdakao-Usansolo
Other Study IDs: PI06/1010; 061017, 06714, 060326, 0664 (Other Grant/Funding Number: Fondo de Investigación Sanitaria); 2012111008 (Other Grant/Funding Number: Departamento de Sanidad del Gobierno Vasco)
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: COPD
Keywords: Chronic Obstructive Pulmonary Disease; Disease Exacerbation Clinical Prediction Rule; Decision Analysis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Objectives: To estimate the rate of appropriate hospital admissions , and of discharge to home episodes that would have been appropriate admissions to the hospital, on patients with exacerbations of their COPD by using appropriateness explicit criteria developed with the RAND appropriateness methodology. To evaluate the validity of those criteria by looking at their correlation with morbid-mortality, use of medications and health resources. To identify the variability in the appropriateness admission/discharge among the different centres participating on the study.

Methodology: Prospective observational cohort study. 1. The investigators will apply the previously developed explicit criteria to a sample of COPD exacerbations presented in each of the Emergency Department of each participating hospital (16 centres). 2. The investigators will evaluate if there is variability among centres by comparing their appropriateness rates. 3. To study the validity of the criteria, on those admitted the investigators will collect information on their evolution (length of stay, need of medication, quality of life), complications, vital status during their admission until discharge, and up to 2 months after the visit to the Emergency Department the vital status, complications, readmissions and quality of life. On those discharged to home from the Emergency Department, the investigators will check the presence of complications, vital status, readmissions and quality of life. People trained will collect all the needed information, in the Emergency Department, during their admission, or by personal interview to all discharged to home and to all at 2 months after the visit to the Emergency Department.

DETAILED DESCRIPTION:
A prospective cohort study was performed to validate the explicit criteria developed by the RAM. Other goals for the cohort study were: to predict mortality, ICU or IRCU admission, hospital length of stay, changes in symptoms and to evaluate variability among hospitals in the appropriateness of hospital admission of patients experiencing COPD exacerbations and to study variability in access to care and outcomes. Sixteen hospitals belonging to the Spanish National Health Service agreed to participate: Hospital Costa del Sol, Hospital Valme, Hospital de Motril, Corporació Sanitaria Parc Taulí, Hospital del Mar, Hospital Universitario de La Princesa, Hospital Universitario Gregorio Marañón, Hospital Universitario La Paz, Hospital de Móstoles, Hospital Marqués de Valdecilla, Hospital Santa Marina, Hospital San Eloy, Hospital Galdakao-Usansolo, Hospital Txagorritxu, Complejo Hospitalario Donostia, and Hospital Cruces.

Patients attending the EDs of any of the 16 hospitals with an exacerbation of COPD were informed of the goals of the study and invited to voluntarily participate in it. All information was kept confidential. The Institutional Review Boards of the participating hospitals approved this project. Recruitment started in June 2008 and ended in September 2010.

Patients were candidates for the study if they presented to the ED of any of the participating hospitals with symptoms consistent of an exacerbation of COPD. Exacerbation was defined as an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough, and/or sputum that was beyond normal day-to-day variations, was acute in onset, and may have warranted a change in regular medication in a patient with underlying COPD. Two possible presentations were considered:

Existing COPD. Patients were considered to have been previously diagnosed with COPD if they had a FEV1/forced vital capacity (FVC) quotient <70%, and a negative bronchodilation test with FEV1 change <200 mL and under 15% of the baseline value.

New COPD. Patients not previously diagnosed with COPD but in whom the disease was suspected were also eligible for inclusion in the study. This included smokers or former smokers of more than 15 packs per year with dyspnea, cough, or expectoration for more than three months per year, and experiencing symptoms resembling a clinical manifestation compatible with COPD exacerbation. The diagnosis had to be confirmed by spirometry within 60 days after the index episode at a time when the patient was stable, i.e., the absence of any increase in symptoms or changes in background therapy. If a diagnosis of COPD was not confirmed, the patient was excluded from the study.

Patients were excluded from the study if they had COPD complicated by a comorbidity such as pneumonia, pneumothorax, or pulmonary embolism; lung cancer; or left cardiac insufficiency. Other exclusion criteria included a diagnosis of asthma, extensive bronchiectasis, sequelae of tuberculosis, pleural thickening, or restrictive diseases. Patients who did not wish to participate were also excluded.

Data collected for the cohort study A substantial amount of clinical and other data were needed to meet the objectives of the IRYSS-CAS. Data from several time points were needed: during the patient's evaluation in the ED; at the time the decision was made to hospitalize the patient or discharge him or her to home; in the medical ward (if needed); and during post-hospitalization or post-discharge follow-up. It must be noted that ED physicians were not asked to gather any information other than what they would usually collect for a patient experiencing an exacerbation of COPD. Instead, trained data managers gathered data from hospital and primary care medical records using a manual of instructions that aimed to standardize data collection.

Some of the information required a review of the patient's medical records. Patients admitted to the hospital were interviewed at 1 and 7 days after admission. Patients discharged from the ED to home were interviewed by telephone at, around, 1 and 7 days after discharge. All patients were interviewed by telephone 60 days after the index event.

In the ED. As is true for almost any encounter in the ED, substantial information is gathered for a patient experiencing an exacerbation of COPD. The main data collected were those related to the patient's respiratory function (gasometry, respiratory rate, dyspnea), consciousness level measured by the Glasgow Coma scale, background, and presence of other pathologies as those recorded in the Charlson Comorbidity Index.

At the time of decision making. Data collected at the ED decision time was related to the patient's respiratory status at that moment as well as variables needed to create the appropriateness scenarios, determine the severity of the exacerbation, and evaluate other study criteria .

In the hospital. For patients admitted to the hospital, we collected data directly from the patient's medical record and from a direct interview with him or her from the first day after admission until discharge. Patients were interviewed about their general health status (response to question 1 of the Short Form 36 (SF-36) questionnaire[16]), degree of dyspnea, based on the Medical Research Council Dyspnea Index[17], physical activity level (based on a scale employed previously in various studies and also completed the EuroQol-5D. Patients were also asked about social support and level of functional dependency. This information was recorded in the first 24 hours after arrival to the ED and at discharge.

Following discharge to home from the ED. Among patients discharged to home from the ED, telephone interviews were conducted around 1 day, 7 days, and 60 days after discharge to assess the level of dyspnea, physical activity, and general health (see previous description), the use of and response to medications, need for supplemental oxygen, the need for visits to the patient's primary care physician, subsequent ED visits or hospital readmissions, vital status, presence of other symptoms, social support, and level of functional dependency.

During follow-up. Data collected during follow-up included general health status (SF-36 question), degree of dyspnea, physical activity level, and quality of life, all as previously described. Readmission within 30 days of the index exacerbation for the same reason, or readmission for any reason between 31 and 60 days after the index exacerbation was recorded, as were complications, including all signs, symptoms, syndromes or diseases, which appeared or worsened during the 60-day observation period attributable to COPD or its treatment. For all patients with known COPD, additional variables collected from medical records include baseline severity of COPD as measured by FEV1; hospital admissions during the previous 12 months; baseline therapy (inhaled long-acting beta agonist, long-acting anticholinergics, inhaled corticosteroid and/or supplemental oxygen), the presence of associated diseases such as diabetes, hypertension, ischemic heart disease and/or valve disease, cor pulmonale, peptic ulcer disease, psychiatric disorders, rheumatic disease, history of stroke or deep vein thrombosis, and others needed to determine the Charlson Comorbidity Index.

Mortality information at one year was also recorded for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for the study if they presented to the Emergency Department with symptoms consistent of an exacerbation COPD. COPD was confirmed if the patient had a forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) quotient <70%. When COPD was newly diagnosed during the Emergency Department visit, to be included in the study a patient had to have COPD confirmed by spirometry within 60 days of the index episode at a time when he or she was stable.

Exclusion Criteria:

* Patients were excluded from the study if, at the time they were seen in the Emergency Department , the exacerbation COPD was complicated by a comorbidity such as pneumonia, pneumothorax, pulmonary embolism, lung cancer, or left cardiac failure. Patients who did not wish to participate were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an exacerbation of chronic obstructive pulmonary disease attending the emergency departments (ED) of 16 hospitals in Spain
Sampling Method: Non-Probability Sample
Enrollment: 2487 (Actual)
Dates: Start 2006-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Appropriateness of hospital admission | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  Appropriateness judgement by specific RAND panel criteria

SECONDARY OUTCOMES:
Readmission | 2 months
  Hospital readmission
Length of hospital stay | Hospital admission
Change in symptoms and HRQoL parameters | Up to 2 months
  Changes in dyspnea, physical activity or EuroQol scores
Mortality data | 30 days; at admission or 7 days; at 2 months; at one year
  Death by any cause, or respiratory cause
Intensive Care Unit admission | Hospital admission
  admission to the intensive care unit, and/or requiring invasive or noninvasive
Intermediate Respiratory Care Unit admission | Hospital admission

REFERENCES:
- [Background] Quintana JM, Esteban C, Barrio I, Garcia-Gutierrez S, Gonzalez N, Arostegui I, Lafuente I, Bare M, Blasco JA, Vidal S; IRYSS-COPD Group. The IRYSS-COPD appropriateness study: objectives, methodology, and description of the prospective cohort. BMC Health Serv Res. 2011 Nov 24;11:322. doi: 10.1186/1472-6963-11-322. PMID 22115318
- [Result] Esteban C, Quintana JM, Garcia-Gutierrez S, Anton-Ladislao A, Gonzalez N, Bare M, Fernandez de Larrea N, Rivas-Ruiz F; IRYSS-COPD group. Determinants of change in physical activity during moderate-to-severe COPD exacerbation. Int J Chron Obstruct Pulmon Dis. 2016 Feb 3;11:251-61. doi: 10.2147/COPD.S79580. eCollection 2016. PMID 26893555
- [Result] Esteban C, Arostegui I, Garcia-Gutierrez S, Gonzalez N, Lafuente I, Bare M, Fernandez de Larrea N, Rivas F, Quintana JM; IRYSS-COPD Group. A decision tree to assess short-term mortality after an emergency department visit for an exacerbation of COPD: a cohort study. Respir Res. 2015 Dec 22;16:151. doi: 10.1186/s12931-015-0313-4. PMID 26695935
- [Result] Garcia-Gutierrez S, Quintana JM, Unzurrunzaga A, Esteban C, Bare M, Fernandez de Larrea N, Pulido E, Rivas P, -Copd Group I. Predictors of Change in Dyspnea Level in Acute Exacerbations of COPD. COPD. 2016 Jun;13(3):303-11. doi: 10.3109/15412555.2015.1078784. Epub 2015 Dec 14. PMID 26667827
- [Result] Pomares X, Monton C, Bare M, Pont M, Estirado C, Gea J, Quintana JM, Vidal S, Santiago A; IRYSS-COPD Appropriateness study group. Emergency Hospital Care for Exacerbation of COPD: Is Inhaled Maintenance Therapy Modified? COPD. 2016;13(1):11-8. doi: 10.3109/15412555.2015.1043517. Epub 2015 Sep 29. PMID 26417965
- [Result] Barrio I, Arostegui I, Rodriguez-Alvarez MX, Quintana JM. A new approach to categorising continuous variables in prediction models: Proposal and validation. Stat Methods Med Res. 2017 Dec;26(6):2586-2602. doi: 10.1177/0962280215601873. Epub 2015 Sep 18. PMID 26384514
- [Result] Rivas-Ruiz F, Redondo M, Gonzalez N, Vidal S, Garcia S, Lafuente I, Bare M, Cano Aguirre Mdel P, Quintana-Lopez JM; Grupo IRYSS-COPD. Appropriateness of diagnostic effort in hospital emergency room attention for episodes of COPD exacerbation. J Eval Clin Pract. 2015 Oct;21(5):848-54. doi: 10.1111/jep.12390. Epub 2015 Jul 2. PMID 26139468
- [Result] Garcia-Gutierrez S, Unzurrunzaga A, Arostegui I, Quintana JM, Pulido E, Gallardo MS, Esteban C; IRYSS-COPD group. The Use of Pulse Oximetry to Determine Hypoxemia in Acute Exacerbations of COPD. COPD. 2015;12(6):613-20. doi: 10.3109/15412555.2014.995291. Epub 2015 Mar 16. PMID 25774875
- [Result] Quintana JM, Esteban C, Unzurrunzaga A, Garcia-Gutierrez S, Gonzalez N, Lafuente I, Bare M, de Larrea NF, Vidal S; IRYSS-COPD Group. Prognostic severity scores for patients with COPD exacerbations attending emergency departments. Int J Tuberc Lung Dis. 2014 Dec;18(12):1415-20. doi: 10.5588/ijtld.14.0312. PMID 25517805
- [Result] Quintana JM, Unzurrunzaga A, Garcia-Gutierrez S, Gonzalez N, Lafuente I, Bare M, de Larrea NF, Rivas F, Esteban C; IRYSS-COPD Group. Predictors of Hospital Length of Stay in Patients with Exacerbations of COPD: A Cohort Study. J Gen Intern Med. 2015 Jun;30(6):824-31. doi: 10.1007/s11606-014-3129-x. Epub 2014 Dec 4. PMID 25472508
- [Result] Quintana JM, Esteban C, Garcia-Gutierrez S, Aguirre U, Gonzalez N, Lafuente I, Bare M, Fernandez de Larrea N, Rivas-Ruiz F; IRYSS-COPD Group. Predictors of hospital admission two months after emergency department evaluation of COPD exacerbation. Respiration. 2014;88(4):298-306. doi: 10.1159/000365996. Epub 2014 Sep 10. PMID 25228470
- [Result] Garcia-Gutierrez S, Quintana JM, Bilbao A, Unzurrunzaga A, Esteban C, Bare M, Giron Moreno RM, Pulido E, Rivas P; IRYSS-COPD Appropriateness Study (IRYSS-COPD) Group. Validity of criteria for hospital admission in exacerbations of COPD. Int J Clin Pract. 2014 Jul;68(7):820-9. doi: 10.1111/ijcp.12397. Epub 2014 Feb 20. PMID 25077290
- [Result] Quintana JM, Esteban C, Unzurrunzaga A, Garcia-Gutierrez S, Gonzalez N, Barrio I, Arostegui I, Lafuente I, Bare M, Fernandez-de-Larrea N, Vidal S; IRYSS-COPD group. Predictive score for mortality in patients with COPD exacerbations attending hospital emergency departments. BMC Med. 2014 Apr 23;12:66. doi: 10.1186/1741-7015-12-66. PMID 24758312
- [Result] Vidal S, Gonzalez N, Barrio I, Rivas-Ruiz F, Bare M, Blasco JA, Ruiz-Frutos C, Quintana JM; Investigacion en Resultados y Servicios Sanitarios (IRYSS) COPD Group. Predictors of hospital admission in exacerbations of chronic obstructive pulmonary disease. Int J Tuberc Lung Dis. 2013 Dec;17(12):1632-7. doi: 10.5588/ijtld.13.0177. PMID 24200281
- [Result] Garcia-Gutierrez S, Quintana JM, Barrio I, Bare M, Fernandez N, Vidal S, Gonzalez N, Lafuente I, Arteta E, Esteban C, Pulido E; IRYSS-COPD Appropriateness Study (IRYSS-CAS) group. Application of appropriateness criteria for hospitalization in COPD exacerbation. Intern Emerg Med. 2013 Jun;8(4):349-57. doi: 10.1007/s11739-013-0927-9. Epub 2013 Mar 19. PMID 23508735
- [Result] Garcia-Gutierrez S, Quintana JM, Aguirre U, Esteban C, Bilbao A, Escobar A, Vidal S, Bare M, Aizpuru F, Blasco JA; Investigacion en Resultados y Servicios Sanitarios (IRYSS) COPD Group. Explicit criteria for hospital admission in exacerbations of chronic obstructive pulmonary disease. Int J Tuberc Lung Dis. 2011 May;15(5):680-6. doi: 10.5588/ijtld.10.0408. PMID 21756522
- [Result] Bare M, Montón C, Pomares X, Font J, Torá N, Estirado C, Quintana JM, Santiago A, Vidal S, The Iryss-COPD appropiateness Study Group. Cohort study of factors contributing to mortality two months after exacerbation of COPD according to patient destination from emergency department. British Journal of Medicine and Medical Research 5(2):221-234, 2015
- [Result] Arostegui I, Esteban C, Garcia-Gutierrez S, Bare M, Fernandez-de-Larrea N, Briones E, Quintana JM; IRYSS-COPD Group. Subtypes of patients experiencing exacerbations of COPD and associations with outcomes. PLoS One. 2014 Jun 3;9(6):e98580. doi: 10.1371/journal.pone.0098580. eCollection 2014. PMID 24892936
- [Result] Barrio I, Arostegui I, Quintana JM, Group IC. Use of generalised additive models to categorise continuous variables in clinical prediction. BMC Med Res Methodol. 2013 Jun 26;13:83. doi: 10.1186/1471-2288-13-83. PMID 23802742
- [Result] García-Gutiérrez S, Quintana JM, Unzurrunzaga A, Esteban C, González N, Barrio I. Creación de una escala para evaluar la gravedad de las exacerbaciones agudas de la enfermedad pulmonar obstructiva crónica (EA-EPOC) en los servicios de urgencias hospitalarios. Emergencias 26: 251-258, 2014.
- [Derived] Arostegui I, Legarreta MJ, Barrio I, Esteban C, Garcia-Gutierrez S, Aguirre U, Quintana JM; IRYSS-COPD Group. A Computer Application to Predict Adverse Events in the Short-Term Evolution of Patients With Exacerbation of Chronic Obstructive Pulmonary Disease. JMIR Med Inform. 2019 Apr 17;7(2):e10773. doi: 10.2196/10773. PMID 30994471